CLINICAL TRIAL: NCT02120716
Title: Computer Intervention for HIV/STI Risk and Drug Use During Pregnancy
Brief Title: The Health Check-Up for Expectant Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Golfo Tzilos, Behavioral Medicine Research, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HD0756658
Record Dates: First submitted 2014-04-15; First posted 2014-04-23 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: HIV
Keywords: HIV; STIs; Health Check Up; Intervention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Check-Up of Expectant Moms (Experimental): Participants receive computer delivered intervention (Health Check-up for Expectant Moms)
  Interventions: Behavioral: Health Check-Up for Expectant Moms
- Time and attention matched control group (No Intervention): Participants will be presented a brief series of videos of television shows, with subsequent ratings of subjective preference

INTERVENTIONS:
Behavioral: Health Check-Up for Expectant Moms — Participants randomly assigned to the treatment condition will receive a 60-minute brief intervention on the Tablet after the baseline assessment. The software will personalize the intervention content based on the current risk status of each participant and will include a plan addressing endorsed risks. Within one month of baseline, there will be a 15-20 minute, computer-delivered booster session reviewing the personalized plan and identifying barriers in the reduction or risks and/or meeting the goals in the plan.
  Arms: Health Check-Up of Expectant Moms

SUMMARY:
The objective of this study is to develop and determine feasibility of a computer-delivered intervention (Health Check-up for Expectant Moms) approach to target women at risk for HIV or other sexually transmitted infections (STIs) and alcohol/drug use during pregnancy through two phases of testing:

The development aims of this study are to:

1. Develop intervention content.
2. Perform a small open trial (n = 10) of the computer based intervention (Health Check-up for Expectant Moms) to assess feasibility of recruitment of target population and acceptability of the intervention and study procedures via participant report of ease of use, helpfulness, and overall satisfaction.

The pilot study aims of this study are to:

1. Conduct a randomized controlled pilot study in a sample of 50 high risk (at risk for HIV/STIs and alcohol/drug use) pregnant women.
2. Determine:

   1. feasibility of the computer based intervention
   2. acceptability via participant report of ease of use, helpfulness, and overall satisfaction
   3. evidence for the hypothesized effects on outcomes: the proposed intervention, in comparison to a time-and-attention-matched control group, will produce reductions in HIV/STIs risk behavior during the follow-up assessment at 4 months.
3. Determine if the intervention condition, relative to control, will produce reductions in alcohol/drug use (frequency, quantity, and heavy drinking/use frequency).
4. Determine effects on process variables: if participants assigned to the intervention condition, relative to control, will demonstrate greater increases in knowledge, readiness to change and risk perceptions.

DETAILED DESCRIPTION:
This R21 will assess a computer-delivered screening, brief intervention and referral to treatment (SBIRT) approach, the Health Check-up for Expectant Moms (HCEM), which will address barriers in early identification and intervention with women at risk for HIV/STI primarily, integrating substance use given the well-supported relationship between these risks during pregnancy. The study will accomplish these objectives by developing and pilot testing a tailored, motivationally enhanced HIV/STI and alcohol/drug use risk reduction intervention that incorporates motivational interviewing (MI) and is consistent with the Information-Motivation-Behavior model of HIV risk behavior. The HCEM is a computer-delivered, brief intervention (one 60-minute session, plus a 15-minute booster session within one month) that is theory-driven and derived from empirical support. The study consists of the following phases: during the Development Phase, the research team will adapt the software for the computer-delivered intervention and an open trial with 10 participants. During the Pilot Study Phase, we will conduct a two-group, randomized controlled study with a sample of 50 pregnant women endorsing HIV/STI and alcohol/drug use risk. Study procedures include the following: potential participants will complete a 10-minute computer-based screener, including questions about general health, alcohol and drug use, and sexual behavior. Inclusion criteria for participation in the study include pregnant women who endorse: 1) an unplanned pregnancy, 2) at least one unprotected vaginal (or anal) sex occasion (USO) in the past 30 days, and 3) current alcohol or drug use, or at risk for prenatal alcohol/drug use. Participants who meet criteria for the study based on the screener will be consented and complete the computer-delivered baseline assessment. Study participants will complete a 60-minute, computer-delivered intervention at baseline, and a 15-minute computer-delivered booster session within one month. Participants will be randomly assigned to either the HCEM (i.e., motivational interviewing-based brief intervention) or a time-and-attention-matched control group (i.e., a brief series of videos of television shows, with subsequent ratings of subjective preference). All participants will complete a computer-delivered, follow-up assessment at four months. Results of this program of research are expected to inform the development of integrated HIV/STI and alcohol/drug use interventions that are high-reaching and widely disseminable within prenatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Are pregnant
2. Endorse having an unplanned pregnancy
3. Endorse at least one unprotected sex occasion (USO) in the past 30 days
4. Endorse current alcohol or drug use or are at-risk for prenatal alcohol/drug use
5. Are between 18 and 50 years old.
6. Are able to speak and read English sufficiently to be able to complete the study procedures.

Exclusion Criteria:

1. Unable to provide informed consent
2. Cannot understand English well enough to understand the consent form when read aloud or assessment instruments that are narrated by the computer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golfo Tzilos, PhD, Principal Investigator — Butler Hospital; Caron Zlotnick, PhD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Tzilos Wernette G, Plegue M, Kahler CW, Sen A, Zlotnick C. A Pilot Randomized Controlled Trial of a Computer-Delivered Brief Intervention for Substance Use and Risky Sex During Pregnancy. J Womens Health (Larchmt). 2018 Jan;27(1):83-92. doi: 10.1089/jwh.2017.6408. Epub 2017 Oct 5. PMID 28981379

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Check-Up of Expectant Moms: Participants receive computer delivered intervention (Health Check-up for Expectant Moms)
  Health Check-Up for Expectant Moms: Participants randomly assigned to the treatment condition will receive a 60-minute brief intervention on the Tablet PC after the baseline assessment. The software will personalize the intervention content based on the current risk status of each participant and will include a plan addressing endorsed risks. Within one month of baseline, there will be a 15-20 minute, computer-delivered booster session reviewing the personalized plan and identifying barriers in the reduction or risks and/or meeting the goals in the plan.
Period: Overall Study
Arm/Group | Health Check-Up of Expectant Moms | Time and Attention Matched Control Group
Started | 31 | 19
Completed | 30 | 19
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Check-Up of Expectant Moms | Time and Attention Matched Control Group | Total
Number analyzed (Participants) | 31 | 19 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.1 (5.79) | 23.2 (4.3) | 24.4 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 19 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 23 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 2 | 13
  White | 7 | 8 | 15
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 31 | 19 | 50

OUTCOME MEASURES:

1. Primary Outcome: CIAS (Computerized Intervention Authoring Software) Satisfaction Measure Scores to Assess the Feasibility and Acceptability of the Computer and HCEM Software
Description: CIAS Satisfaction Measure (adapted from Ondersma et al., 2005). Self-report instrument assessing the extent to which participants found the software acceptable. Mean ratings on items including Likeability and Ease of use; scores range from 1 (low) to 5 (high) in satisfaction.
  HCEM Satisfaction Measure. Self-report instrument assessing the extent to which participants found specific components of the HCEM intervention acceptable (e.g., videos, resources, information); scores range from 1 (low) to 7 (high) in satisfaction.
Time Frame: 4 month follow up
Population: Participants in the HCEM (intervention) condition reported on their satisfaction with the computer software and specific HCEM intervention components.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Health Check-Up of Expectant Moms
Number analyzed (Participants) | 31
units on a scale
  CIAS measure | 4.8 [4.6 to 5.0]
  HCEM measure | 6.6 [6.3 to 6.8]

2. Secondary Outcome: Percentage of Participants With Reduced HIV/STI Risk Behavior (Condomless Sex) From Baseline to Follow-Up.
Description: Participants completed the Timeline Followback interview and self-reported their daily sex risk behavior including condomless sex
Time Frame: 4 month follow up
Measure: Number; unit: percentage of participants
Arm/Group | Health Check-Up of Expectant Moms | Time and Attention Matched Control Group
Number analyzed (Participants) | 31 | 19
percentage of participants | 27 | 5
Statistical Analysis 1: Comparison: Health Check-Up of Expectant Moms; Test type: Other — Logistic regression analysis; p = 0.13, Regression, Logistic; Odds Ratio (OR) = 5.5, 95% CI 2-sided [0.6 to 51.2]

3. Secondary Outcome: Percentage of Participants Endorsing Alcohol/Drug Use at Baseline and 4-Month Follow-Up
Description: The Timeline Followback approach was used to collect self-reported data regarding alcohol and/or drug use over a 4-month time period.
Time Frame: Baseline and 4-Month Follow-Up
Population: The clustering within subject was accounted for using a generalized estimating equations (GEE) approach.
Measure: Number; unit: percentage of participants
Arm/Group | Health Check-Up of Expectant Moms | Time and Attention Matched Control Group
Number analyzed (Participants) | 31 | 19
percentage of participants
  Baseline assessment | 77 | 58
  Follow-up assessment | 23 | 42
Statistical Analysis 1: Comparison: Time and Attention Matched Control Group; The reported percentages were captured at two separate time points (baseline, and at 4-Month Follow-Up); Test type: Superiority; p < 0.015, Regression, Logistic; Odds Ratio (OR) = 11.7, 95% CI 2-sided [4.2 to 33.0]

ADVERSE EVENTS:
Arm/Group | Health Check-Up of Expectant Moms | Time and Attention Matched Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/19
Serious Adverse Events (participants affected / at risk) | 5/31 | 1/19
Other Adverse Events (participants affected / at risk) | 0/31 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Check-Up of Expectant Moms (N=31) | Time and Attention Matched Control Group (N=19)
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Partner violence (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Participant reported she was "kicked in the stomach" by her partner. Had routine medical visit and reported no medical complications as a result of incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No